CLINICAL TRIAL: NCT07156409
Title: A Prospective, Multicenter, Single-Arm Target Value Study Evaluating the Safety and Effectiveness of a Peripheral Embolization Coil System for the Treatment of Arteriovenous Embolization in the Peripheral Vasculature in a Real-World Setting
Brief Title: The Clinical Application of Peripheral Embolization Coil Systems in Arteriovenous Embolization Within the Peripheral Vasculature
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Zenith Vascular Scitech Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZTHTL202501
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Arterial Hemorrhage; Arteriovenous Malformation; Arteriovenous Fistula; Peripheral Aneurysm
MeSH Terms: conditions — Arteriovenous Malformations; Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peripheral Embolization Coil System (Experimental)
  Interventions: Device: Peripheral Embolization Coil System

INTERVENTIONS:
Device: Peripheral Embolization Coil System — Primarily used to block or reduce the blood flow velocity in the peripheral vascular system

SUMMARY:
Evaluation of the Safety and Effectiveness of the Peripheral Embolization Coil System Manufactured by Suzhou Zhongtian Medical Instruments Co., Ltd. for the Treatment of Arteriovenous Embolization in the Peripheral Vasculature in a Real-World Setting

DETAILED DESCRIPTION:
This study adopts a prospective, multicenter, single-arm target value design. It plans to enroll patients with peripheral arteriovenous diseases requiring embolization, who will be treated using the Peripheral Embolization Coil System manufactured by Suzhou Zhongtian Medical Instruments Co., Ltd. Follow-up assessments will be conducted during the procedure, prior to discharge, and at 30 days, 3 months, and 6 months post-operation to evaluate the safety and effectiveness of the Peripheral Embolization Coil System

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years (inclusive), regardless of gender;
2. Patients diagnosed preoperatively via imaging (including but not limited to ultrasound, CTA, MRA, DSA, etc.) with peripheral arteriovenous conditions requiring embolization therapy;
3. The visually estimated normal reference diameter of the target vessel is ≥ 3mm;
4. Patients or their legally authorized representatives are capable of understanding the study objectives, voluntarily participating in this study, providing signed informed consent, and able to comply with follow-up.

Exclusion Criteria:

1. The target vessel requires the concurrent use of other embolic materials (e.g., Gelfoam, embolic microspheres, liquid embolic agents, etc.);
2. Known definite history of allergy to platinum, tungsten metals, and/or any component of the investigational product;
3. Subjects with pre-existing severe cardiac, hepatic, renal, respiratory diseases, or coagulation disorders who are unsuitable for anesthesia or endovascular surgical treatment;
4. High-flow arteriovenous fistulas that may cause migration of the embolic material;
5. The target aneurysm is a blister aneurysm, dissecting aneurysm, mycotic (infectious) aneurysm, ruptured aneurysm, or aneurysm caused by connective tissue diseases;
6. Severe vascular stenosis or tortuosity, or anatomical anomalies where it is anticipated that the device will be difficult to navigate to the lesion site, or other uncommon anatomies that may interfere with device use;
7. The target vessel has undergone any previous embolization therapy or surgical intervention, or has recurrent disease;
8. Definite allergy, resistance, or contraindication to antiplatelet drugs, anticoagulants, contrast media, and/or anesthetics;
9. Females who are pregnant, breastfeeding, or planning to become pregnant within 6 months; males planning for parenthood within the next 6 months;
10. Subjects currently participating in other drug or device clinical trials who have not reached the trial endpoint;
11. Investigators deem the subject unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of technical success (embolization of target vessel) | Immediately after the intervention
  Angiographic imaging confirmed successful occlusion of the target vessel segment with no blood perfusion.

SECONDARY OUTCOMES:
Rate of treated vessel occlusion | 6 months
  Angiographic imaging confirmed successful occlusion of the target vessel segment with no blood perfusion.
Target Vessel Re-intervention Rate | 30 days,3 months,6 months from procedure date
  The embolized segment of the target vessel requires re-intervention/surgical intervention.
All-cause mortality rate | 6 months from procedure date
  Death from any cause
Rate of Device/Procedure-Related Serious Adverse Events | Perioperative,30 days,3 months,6 months from procedure date
Adverse Event/Serious Adverse Event Rate | 6 months from procedure date